CLINICAL TRIAL: NCT05013190
Title: Clinical Outcome of Ixazomib (NINLARO®) Based Regimens in Chinese Patients With Multiple Myeloma Previously Receiving a Bortezomib/Carfilzomib-Based (re)Induction Regimen in Clinical Setting of Real World: An Open-Label, Single-Arm, Multicenter, Observation Study
Brief Title: A Study of NINLARO® in Chinese Adults With Multiple Myeloma
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C15058
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Multiple Myeloma (MM): Participants diagnosed with MM (newly diagnosed multiple myeloma [NDMM] and first relapse multiple myeloma [FRMM]) using International Myeloma Working Group (IMWG) criteria who received a bortezomib/carfilzomib-based triple-drug regimens for more than 2 cycles as initial therapy, achieved at least partial response (PR) as defined by IMWG criteria, and are ready to start receiving an ixazomib containing therapy prescribed by their treating physician will be observed prospectively for 24 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to check side effects and results in adults with multiple myeloma after switching from a bortezomib/carfilzomib -based to an Ixazomib-based treatment.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with multiple myeloma (MM). Participants will be treated with ixazomib based regimens until progression or unacceptable toxicity leading to a discontinuation or change in regimen, for a maximum of 26 cycles (24 months) (as per NINLARO® label) in real world clinical setting.

The study will enroll approximately 80 participants. The data will be collected prospectively in medical charts and will be recorded into electronic case report forms (eCRFs). All the participants will be assigned to a single observational cohort:

• Participants with MM

This multi-center trial will be conducted in China. The overall time for data collection in the study will be 24 months. Participants will be followed once every 3 months for a period not exceeding 24 months, ending 12 months after the last participant's enrollment unless withdraw of informed consent form, death or lost to follow-up, termination of the study by the sponsor, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Who was first diagnosed or first relapse MM participants using IMWG 2016 criteria.
2. Diagnosed with multiple myeloma using IMWG 2016 criteria and must be transplant ineligible as determined by their physician, or if transplant eligible, not expect to undergo transplant for at least 24 months after study enrollment.

   a. Stem cell harvest and mobilization regimen is acceptable if clinically indicated. But must first be confirmed by the Takeda Medical Monitor.
3. Who received bortezomib/carfilzomib-based triple-drug regimens as frontline treatment, including bortezomib+cyclophosphamide+dexamethasone (VCD), bortezomib+lenalidomide dexamethasone (VRD), bortezomib+doxorubicin+dexamethasone (PAD), bortezomib+thalidomide+dexamethasone (VTD), bortezomib+pomadomide+dexamethasone (VPD), or carfilzomib+lenalidomide+dexamethasone (KRD), carfilzomib+thalidomide+dexamethasone (KTD), carfilzomib+pomalidomide+dexamethasone (KPD).
4. Must achieve at least partial response (PR) as defined by IMWG criteria after bortezomib/carfilzomib-based initial therapy.
5. Eastern Cooperative Oncology Group (ECOG) 0-2.

Exclusion Criteria:

1. Received a bortezomib/carfilzomib-based triple-drug regimens as initial therapy less than 2 cycles.
2. Failure to have fully recovered (that is, less than or equal to [<=] Grade 1 toxicity) from the reversible effects of prior chemotherapy.
3. Have documented diagnosis of other cancers prior to the diagnosis of MM, excluding squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, which is considered cured with minimal risk of recurrence within 3 years.
4. Has >=Grade 2 peripheral neuropathy (PN), or Grade 1 with pain on clinical examination at the time of enrollment.
5. Previously been treated with ixazomib or participated in a study with ixazomib whether treated with ixazomib or not.
6. Have gastrointestinal (GI) disease or procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
7. Have an active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been first diagnosed with MM and FRMM using IMWG criteria, and who have received a bortezomib/carfilzomib-based triple-drug regimens (more than 2 cycles) as initial therapy, and must achieve at least PR as defined by IMWG criteria at the time of enrollment will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) at 24 Months | From the date of first administration of ixazomib therapy to the date of first documentation of PD or death, lost to follow-up, whichever occurs first (up to 24 months)
  PFS:time date of first administration of ixazomib therapy to date of first documentation of progressive disease(PD)/death,lost to follow-up,whichever occurs first as per IMWG 2016 Response Criteria.PD:increase of 25 percent(%) from lowest confirmed response value in any one/more of following:Serum and Urine M-protein only in participants without measurable serum and urine M-protein levels,difference between involved/uninvolved free light chain (FLC) levels(absolute increase greater than(>)10 milligram per deciliter [mg/dL]),and without measurable involved FLC levels, bone marrow plasma-cell% irrespective of baseline status (absolute increase must be ≥10%); appearance of new lesions, ≥50% increase from nadir in SPD of >1 lesion/ ≥50% increase in the longest diameter of a previous lesion >1 centimeter in short axis; ≥50% increase in circulating plasma cells (minimum of 200 cells per microliter [mcL]) if this is the only measure of disease. It will be analyzed using Kaplan-Meier method.

SECONDARY OUTCOMES:
Time to Next Treatment (TTNT) | From the date of the first administration of ixazomib therapy to first dose of new treatment (up to 24 months)
  Time to next treatment will be defined as the time from the date of the first administration of ixazomib therapy to first dose of new treatment given after changing the therapy.
Percentage of Participants Achieving Very Good Partial Response (VGPR) | Up to 24 months
  VGPR will be assessed as per IMWG 2016 Response Criteria, and defined as: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or greater than or equal to (>=) 90% reduction in serum M-protein plus urine M-protein level less than (<) 100 milligram (mg) per 24 hour (h).
Percentage of Participants Achieving Complete Response (CR) | Up to 24 months
  CR will be assessed as per IMWG 2016 Response Criteria and defined as: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. For participants who only rely on serum FLC level as measurable lesions, in addition to meeting the above CR criteria, the ratio of serum FLC should return to normal under two consecutive assessments.
Percentage of Participants Achieving Stringent Complete Response (sCR) | Up to 24 months
  sCR will be assessed as per IMWG 2016 Response Criteria, and defined as: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. For participants who only rely on serum FLC level as measurable lesions, in addition to meeting the above CR criteria, the ratio of serum FLC should return to normal under two consecutive assessments. Absence of clonal plasma cells in bone marrow biopsy by immunohistochemistry. Presence of bone clonal plasma cells is defined as κ/λ >4:1 or <1:2 ratio under two consecutive detection by immunohistochemical method (for participants with type κ and type λ respectively, and requiring a minimum of 100 plasma cells for analysis).
Duration of Ixazomib Therapy (DOT) | Up to 24 months
  DOT will be defined as the time from the date of the first administration of ixazomib therapy to the date of the last administration of ixazomib therapy.
Duration of CR | Up to 24 months
  Duration of CR will be defined as time from first documented CR to the date of PD as per IMWG 2016 Response Criteria.
Overall Survival (OS) | Up to 24 months
  OS will be defined as the time from enrollment to death from any cause.
Health-related Quality of Life (HRQOL) Based on European Organization for Research and Treatment of Cancer Multiple Myeloma Module (EORTC QLQ-MY20) | Up to 24 months
  EORTC QLQ-MY20 is self-administered patient-reported outcomes (PRO) used to assess quality of life during the last 7 days. It has 20 items evaluated on 4 point rating scale ranging from: 1 (not at all), 2 (a little), 3 (quite a bit), 4 (very much). Total score ranges from 20 to 80. Higher scores represent worsening.
HRQOL Based on EORTC QLQ-C30 | Up to 24 months
  EORTC QLQ-C30 is self-administered PRO which contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/quality of life (QOL) scale. EORTC QLQ-C30 contains 28 questions (4-point scale where 1=Not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=Very poor [worst] to 7= Excellent [best]). Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QOL scale, higher scores represent better QOL; for the symptom scales, lower scores represent better QOL.
Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Up to 24 months
  TSQM-9 is self-administered PRO. It is a 9-item, validated, self-administered instrument used to assess participant's satisfaction or dissatisfaction with medication. The three domains assessed are effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain.
Number of Participants Categorized Based on Healthcare Resource Utilization | Up to 24 months
  Healthcare resource utilization will include outpatient visits to the study site, overnight hospital admissions, emergency department visits, and hospice care.
Number of Participants Categorized Based on Reason for Dose Reduction of Ixazomib Therapy | Up to 24 months
Number of Participants Categorized Based on Reason for Interruption of Ixazomib Therapy | Up to 24 months
Number of Participants Categorized Based on Reason for Discontinuation of Ixazomib Therapy | Up to 24 months
Relative Dose Intensity (RDI) | Up to 24 months
  RDI is defined as 100*(Total amount of dose taken)/(Total prescribed dose of treated cycles), where total prescribed dose equals (dose prescribed at enrollment* number of prescribed doses per cycle* the number of treated cycles).
Number of Participants who Experience at Least one Adverse Event (AE) | Up to 24 months
Number of Participants Categorized Based on Occurrence of Second Primary Malignancies (SPM) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- China (12):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Beijing Chao-Yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Henan Province People Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhenzhou University, Zhengzhou, Henan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Qingdao
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Chen W, Liu A, Li L. The MODIFY Study Protocol: An Open-Label, Single-Arm, Multicenter, Prospective Pragmatic Study of Ixazomib-Based Triple-Drug Therapy in Chinese Patients with Multiple Myeloma. Adv Ther. 2023 Feb;40(2):705-717. doi: 10.1007/s12325-022-02355-3. Epub 2022 Dec 4. PMID 36463561
- See also: To obtain more information on the study, click on this link. — https://clinicaltrials.takeda.com/study-detail/611fce65ca0ce2002ab9e659